CLINICAL TRIAL: NCT07307001
Title: Vojta Therapy Versus Conservative Therapy for Patients With Ischemic Stroke in Regaining Functional Independence
Brief Title: Vojta Therapy Versus Conservative Therapy for Patients With Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lucaci Doru Nicolae (Other)
Responsible Party: Sponsor-Investigator, Lucaci Doru Nicolae, Physiotherapist, President Premium Medcenter
Organization: President Premium Medcenter (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 85/22.05.2025
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke | interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): The physiotherapists will apply only the Conservative Therapy to the subjects in this group
  Interventions: Procedure: Conservative therapy
- Study Group (Experimental): The physiotherapists will apply the Conservative Therapy, and in addition will also apply the Vojta Therapy
  Interventions: Procedure: Vojta therapy; Procedure: Conservative therapy

INTERVENTIONS:
Procedure: Vojta therapy — The physiotherapists will apply the techniques and methods of Vojta therapy along with the classical tools of the Conservative therapy. Through the therapeutic use of reflex locomotion involved in Vojta sessions, it can succeed in elementary movement models, meaning that they can be accessible again for patients with central nervous system and musculoskeletal affections.
  Arms: Study Group
Procedure: Conservative therapy — The physiotherapists will apply only the classical tools and methods involved in the Conservative therapy (Bobath, massage, electrotherapy, hydrotherapy).

SUMMARY:
Main hypothesis: Vojta Therapy shows significantly better results in regaining functional independence for patients with ischemic stroke than the Conservative Therapy

The present study wishes to bring evidence that Vojta Therapy is superior in regaining functional independence for patients with ischemic stroke, whether it is solely used in the intervention, or as a complementary tool along with the Conservative Therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients post-ischemic stroke
* patients who meet the age criteria
* patients who have had the stroke in less than 3 years ago

Exclusion Criteria:

* patients with hemoragic stroke
* patients with comorbidities
* noncooperative patients

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Trunk Control Test (TCT) | From enrollment to the end of treatment at 2 weeks, and a follow up at 3 months
  The Trunk Control Test (TCT) will be used to assess the motor function and control of the trunk in participants. The scale contains 5 task-items, each of them being scored between 0 (unable, needs help), 12 (able but abnormal), or 25 (able, normal). The scoring interval is 0-100, where 100 signify better trunk function, and 0 none.
Functional Independence Measure (FIM) | From enrollment to the end of treatment at 2 weeks, and a follow-up at 3 months
  The Functional Independence Measure (FIM) will be used to assess the level of a participant's functional independence in activities of daily living. The test comprises in 18 items, each of which is assigned against a seven-point ordinal scale, where the higher the score for an item, the more independently the patient is able to perform the tasks assessed by that item. Total scores range from 18 to 126.

SECONDARY OUTCOMES:
Trunk Impairment Scale (TIS) | From enrollment to the end of the treatment at 2 weeks, and a follow-up at 3 months
  The Trunk Impairment Scale (TIS) aims to evaluate the trunk in patients who have suffered a stroke. The scale contains 3 subscales (static, dynamic and coordonation), totalling a number of 17 items. The total score varies from 0 to 23, 0 meaning worse trunk control, and 23 best trunk control.
Postural Assessment Scale for Stroke (PASS) | From enrollment to the end of the treatment at 2 weeks, and a follow-up at 3 months.
  The PASS scale is used to measure balance and postural control in stroke survivors across lying, sitting and standing positions. The scale contains 3 subscales (lying, sitting, standing), and 12 tasks, with a total score varying between 0 (worse posture) and 36 (better posture).
Berg Balance Scale (BBS) | From enrollment to the end of the treatment at 2 weeks, and a follow-up at 3 months.
  The BBS scale is used to objectively determine a patient's ability to safely balance during a series of predetermined tasks. The scale contains 14 standardized tasks, scored from 0 (unable), to 4 (independent) for a total of 56 points.
Barthel Index | From enrollment to the end of the treatment at 2 weeks, and a follow-up at 3 months.
  The Barthel Index scale is an ordinal scale which measures a person's ability to complete ADL. The scale evaluates performance in 10 areas, with scores of 0, 5, or 10 for each item. A total score of 0 means total dependence, while 100 means independent.
Nottingham Extended ADL | From enrollment to the end of the treatment at 2 weeks, and a follow-up at 3 months.
  The NEADL scale is a self-report questionnaire used in rehabilitation especially post-stroke, to measure independence in broader daily tasks beyond basic ones. It scores independence on a scale (0-1 or 0-2 points per item, total max 22) with higher scores indicating greater independence. The scale contains 22 items.
Functional Ambulation Categories (FAC) | From enrollment to the end of the treatment at 2 weeks, and a follow-up at 3 months.
  The FAC scale is a 6 point (0-nonfunctional ambulator; 5-ambulator/independent) functional walking test that evaluates ambulation ability, determining how much human support the patient requires when walking. It is not a multi-item questionnaire.
Rivermead Mobility Index (RMI) | From enrollment to the end of the treatment at 2 weeks, and a follow-up at 3 months.
  The RMI scale is a quick tool assessing 15 activities, like turning in bed, sitting balance, transfers, etc. often after stroke/head injury. Scoring varies between 0 (unable) and 1 (able), with a maximum score of 15, higher scores indicating better mobility.
Wisconsin Gait Scale (WGS) | From enrollment to the end of the treatment at 2 weeks, and a follow-up at 3 months.
  The WGS scale is used to monitor the effectiveness of rehabilitation training and the gate problems experienced by the patients after a stroke. With a number of 14 items, the test is generally scored between 1 (normal) and 3 (atypical), with the gait aid item scored 1-5, and knee flexion scored 1-4.

OTHER OUTCOMES:
Stroke Impact Scale (SIS) | From enrollment to the end of the treatment at 2 weeks, and a follow-up at 3 months.
  The SIS scale is a patient-reported outcome measure that evaluates the biopsychosocial aspects of life after stroke. The scale contains 59 items regarding daily acitivites, on a 5-point scale for each item, a greater score meaning less dificulty.
EuroQol-5 Dimension (EQ-5D) | From enrollment to the end of the treatment at 2 weeks, and a follow-up at 3 months.
  The EQ-5D scale is a widely used health questionnaire assessing health-related quality of life, focusing on 5 key areas, with a visual analog scale (VAS). The test contains only 5 items regarding 5 the 5 areas. Scoring for this test is a 5 digit generated code, that is converted into a single utility score (0=death, 1=perfect health).
Stroke Specific Quality of Life (SS-QoL) | From enrollment to the end of the treatment at 2 weeks, and a follow-up at 3 months.
  The SS-QoL scale is a patient-reported tool for assessing health related quality of life in stroke survivors, measuring impacts on daily function, emotions, social roles, and cognition across 12 key domains and 49 items. Scoring for this test varies between 49-245, each item being scored between 1 (total help) and 5 (no help needed).

CONTACTS AND LOCATIONS:
Overall Officials: Doru Nicolae Lucaci, PhD, Principal Investigator — Auxologico President
Locations (1):
- Auxologico President Recovery Hospital, Cordău, Romania

IPD SHARING:
Plan to Share IPD: No
The patient's personal details are strictly confidential. Only the demographic data will be available.